CLINICAL TRIAL: NCT05687188
Title: Evaluating Obesity-Mediated Mechanisms of Pancreatic Carcinogenesis in Minority Populations
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MCC-21962; PA210192, W81XWH2211021 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; biomarkers; health disparities
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Retrospective chart review and sample analysis of both pathologically confirmed Pancreatic Ductal Adenocarcinoma (PDAC) cases and non-Cancer control cases.
- Prospective Cohort: Blood samples, tissue samples and data will be collected from all participants as applicable.
  Interventions: Other: Blood Sample Collection; Other: Tissue Sample Collection; Other: Data Collection; Other: Medical Image Collection

INTERVENTIONS:
Other: Blood Sample Collection — Participants will have 40 mL of blood drawn at baseline/pre-treatment. The study team will aim to have this blood collected at the time of standard of care blood draw if possible.
  Groups: Prospective Cohort
Other: Tissue Sample Collection — At the time of tissue biopsy or surgical resection (if applicable) pancreatic tumor tissue, fat, tissue from site of metastasis, and cyst fluid (if applicable) will be collected.
  Groups: Prospective Cohort
Other: Data Collection — Participants will complete a study questionnaire at baseline that includes medical history, lifestyle, and family history information.
  Groups: Prospective Cohort
Other: Medical Image Collection — Medical images that are obtained during routine care such as computed tomography (CT) scans, magnetic resonance imaging (MRIs) and ultrasounds will be reviewed by the study team throughout the participant's medical care.
  Groups: Prospective Cohort

SUMMARY:
This study will evaluate obesity-mediated mechanisms of pancreatic carcinogenesis in minority populations.

DETAILED DESCRIPTION:
This observational study will evaluate obesity-mediated mechanisms of pancreatic carcinogenesis in minority populations consisting of adult males or females, 18 years of age or older, who self-report as African American (AA) or Non-Hispanic White (NHW), and present to the gastrointestinal (GI) clinic, surgery, or endoscopy at a participating Florida Pancreas Collaborative (FPC) site or University of Mississippi Medical Center (UMMC) with a clinical suspicion or diagnosis of a pancreatic tumor. This study will also include patients who have been previously recruited as part of the FPC study. Our central hypothesis is that adipose tissue (AT) dysfunction contributes to malignant transformation, therapeutic resistance, and poor survival among obese AA pancreatic ductal adenocarcinoma (PDAC) cases and such dysfunction will be characterized by unique biology. The primary objective of this multi-institutional and multidisciplinary translational study is to identify a molecular and imaging profile unique to paired PDAC tumors and AT from AA and harness biological observations to predict therapeutic response and target novel obesity-mediated mechanisms of PDAC development and progression using in vitro, ex vivo, and in vivo techniques and new combinations of drug agents.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older at time of signing informed consent
* Patients who self-report as African American, Non-Hispanic White
* Patients who present to the gastrointestinal (GI) clinic, surgery, or endoscopy at a participating Florida Pancreas Collaborative (FPC) site or the University of Mississippi Medical Center (UMMC) with a clinical suspicion or diagnosis of a pancreatic tumor.

Exclusion Criteria:

* Patient under 18 years of age
* Has no suspicion or diagnosis of a pancreatic cancer or tumor
* Self-reported race/ethnicity other than African American or Non-Hispanic White.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at a Florida Pancreas Collaborative site who identify as African American or Non-Hispanic White.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assess molecular and radiological landscape of traditional PDAC tumors in the context of Race/Ethnicity | at 36 months
  Investigators will compare gene prevalence, type and expression of genetic mutations and radiomic features in African American participants vs Non-Hispanic White participants
Compare biological properties of Adipose Tissue dysfunction | at 36 months
  Investigators will compare biological properties of Adipose Tissue dysfunction between African American vs Non-Hispanic White participants.
Examine the role of Adipose Tissue and PDAC tumor interactions in influencing tumor growth, metastasis, and therapeutic response | at 36 months
  Investigators will compare the biological interactions of Adipose Tissue and PDAC tumor growth between African American vs. Non-Hispanic White participants to develop new and/or targeted drug combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Permuth, PhD, MS, Principal Investigator — Moffitt Cancer Center; Mokenge Malafa, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: Undecided